CLINICAL TRIAL: NCT01665014
Title: Efficacy and Safety of Double Autologous Hematopoietic Stem Cell Transplantation With Sequential Use of Total Marrow Irradiation and High-dose Melphalan in Multiple Myeloma
Brief Title: Total Marrow Irradiation and High-dose Melphalan for Double Autologous Hematopoietic Stem Cell Transplantation in Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMI MM1
Record Dates: First submitted 2012-08-11; First posted 2012-08-15 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Multiple Myeloma
Keywords: autologous hematopoietic stem cell transplantation; total marrow irradiation; melphalan; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Total marrow irradiation (Experimental): Double autologous hematopoietic stem cell transplantation using TMI and HD-Mel
  Interventions: Radiation: Total marrow irradiation

INTERVENTIONS:
Radiation: Total marrow irradiation — Mobilization of stem cells with the use of cytarabine 1.6 g/m2 followed by filgrastim 480 ug/d. Conditioning for the 1st autoHSCT: total marrow irradiation 4 Gy on days -3,-2,-1 (total 12 Gy). Conditioning for 2nd autoHSCT performed 3-4 months after the 1st one: melphalan 100 mg/m2 on days -2,-3 (total 200 mg/m2)

SUMMARY:
The purpose of this study is to evaluate if the use total marrow irradiation (TMI) as a sole preparation for the first autologous hematopoietic stem cell transplantation (autoHSCT) followed by high-dose melphalan used prior to second autoHSCT is safe and effective in patients with multiple myeloma (MM).

DETAILED DESCRIPTION:
AutoHSCT is a standard treatment of patients with MM. According to soem clinical evidence double autoHSCT provides survival advantage compared to a single procedure. Most frequently used conditioning regimen consists pf high doses of melphalan (HD-MEL). In some studies it was used in combination with total body irradiation (TBI), which, however was associated with significant toxicity. In our center the standard procedure includes TBI as a single treatment at 1st autoHSCT and HD-Mel at 2nd autoHSCT.

As in MM malignant plasma cells are localized almost exclusively in bone marrow there is rationale to limit irradiation to bones. For this purpose in the current study we substitute TBI with TMI. Additional boosts are provided for active sites of disease based on PET/CT imaging. Our intention is to minimize toxicity while maintaining the treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Diagnosis of multiple myeloma
* PR, VGPR or CR at inclusion
* Performance status WHO 0-1
* Written informed consent

Exclusion Criteria:

* Organ dysfunction: elevated ALT, AST, bilirubin, AF; creatinine >1.5 upper normal limit; LVEF <45%
* Active infection
* Unstable diabetes
* Psychiatric diseases
* History of high-dose chemotherapy or irradiation
* Second malignancy
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | three years

SECONDARY OUTCOMES:
Rate of complete and very good partial responses | six months

OTHER OUTCOMES:
Rate of severe adverse events | one year

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Giebel, MD, Principal Investigator — Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice Branch, Gliwice, Poland
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice Branch, Gliwice, Poland

REFERENCES:
- [Background] Somlo G, Spielberger R, Frankel P, Karanes C, Krishnan A, Parker P, Popplewell L, Sahebi F, Kogut N, Snyder D, Liu A, Schultheiss T, Forman S, Wong JY. Total marrow irradiation: a new ablative regimen as part of tandem autologous stem cell transplantation for patients with multiple myeloma. Clin Cancer Res. 2011 Jan 1;17(1):174-82. doi: 10.1158/1078-0432.CCR-10-1912. Epub 2010 Nov 3. PMID 21047977